CLINICAL TRIAL: NCT00891800
Title: A Phase II Feasibility Study to Assess the Use of SIR-Sphere in Patients With Breast Cancer Who Have Chemotherapy-Resistant Disease in the Liver
Brief Title: Brachytherapy Radiation Directly to the Liver in Breast Cancer Patients With Metastatic to Liver
Acronym: SIRT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of study patients
Sponsor: St. Joseph's Hospital, Florida (Other)
Responsible Party: Alison Calkins, MD, St. Joseph's Hospital Tampa FL
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJCI023; IDE # G050256
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer Metastatic to the Liver
Keywords: Cancer; Breast; Liver
MeSH Terms: conditions — Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All patients will be treated with SIR-Sphere therapy.
  Interventions: Device: Brachytherapy; Device: SIR-Sphere

INTERVENTIONS:
Device: Brachytherapy — SIR-Sphere contains radiation of Y-90.
  Other Names: Radiation seeds
Device: SIR-Sphere — Brachytherapy Radiation seeds

SUMMARY:
The purpose of this study to study whether or not the use of direct radiation therapy with Y-90 microspheres (SIR-Spheres) has any effect on treated liver with respect to tumor response in breast cancer patients.

Criteria:

* Breast cancer
* Clinical evidence of metastatic disease in the liver
* Performance status (0-2)
* Not pregnant
* Laboratory values received after any prior chemotherapy
* Normal Pt/PTT
* recovered from any chemotherapy side-effects
* No prior radiation therapy to the liver
* No other MAJOR site of cancer such as lungs or brain
* No uncontrolled infections
* a candidate for surgical resection or ablation therapy

DETAILED DESCRIPTION:
Patient must pass an MAA angiography study to detect abnormal shunting of the vessels to the lungs and stomach. Shunting of the radiation seeds to these areas, if an abnormality exists would be harmful.

ELIGIBILITY:
Inclusion Criteria:

* Documented breast cancer
* Clinical evidence of mets to the liver
* Performance status of 0-2
* Life expectancy of greater equal to 3 months
* Not pregnant
* 4 weeks or more since last radiation therapy
* Recovered from all side effects of prior chemotherapy
* Not needing concurrent chemotherapy
* recovered laboratory values
* Bilirubin < 2.0

Exclusion Criteria:

* Candidate for surgical resection or ablation of liver lesion/s
* Prior radiation therapy to the liver
* Co-Morbid disease
* pulmonary insufficiency
* Portal vein thrombosis
* Contraindications to angiography
* > 20 % lung shunting on MAA
* Diffuse extra-hepatic disease
* Concurrent chemotherapy OR capecitabine with 8 weeks
* Failed MAA
* Uncontrolled active infection
* Severe liver dysfunction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Primary: Assessment of the feasibility of SIRT treatment as measured by tumor response in the treated labe/s of the liver.Assessed by CT scan and measurement Secondary Response: Assessment of treatment toxicity. Assessed by examination and blood work. | Patients will be followed for 5 years or Progressive disease in the treated liver or until such time as systemic therapy is needed for disease in other organs which will affect tumor response in the liver.

CONTACTS AND LOCATIONS:
Overall Officials: ALison R Calkins, MD, Principal Investigator — St. Joseph's Hospital, Department of Radiation Therapy
Locations (1):
- St. Joseph's Hospital, Department of Radiation Therapy, Tampa, Florida, United States